CLINICAL TRIAL: NCT06300320
Title: A Randomized, Open-label, Multicenter Phase II Clinical Trial of Rovadicitinib in the Treatment of Third-line and Subsequent Moderate to Severe Chronic Graft-versus-host Disease (cGVHD).
Brief Title: A Clinical Trial of TQ05105 Tablets in the Treatment of Chronic Graft-versus-host Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ05105-II-06
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-11

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ05105 Tablets (Experimental): TQ05105 Tablets administered twice-daily. 28 days as a treatment cycle.
  Interventions: Drug: TQ05105 tablets

INTERVENTIONS:
Drug: TQ05105 tablets — Rovadicitinib (TQ05105) is a novel, oral dual JAK 1/2 and Rho-associated kinases (ROCK) 1/2 inhibitor targeting inflammatory and fibrotic components of cGVHD.

SUMMARY:
This is an open, multi-center clinical study designed to evaluate the efficacy and safety of TQ05105 Tablets in patients with chronic graft-versus-host disease

ELIGIBILITY:
Inclusion Criteria:

* Voluntary and signed informed consent, good compliance;
* Age 18-70 years old; Karnofsky Performance Scale (KPS) ≥60 points; Life expectancy ≥ 6months.
* Received allogeneic hematopoietic stem cell transplantation;
* Diagnosis of moderate-to-severe chronic graft-versus-host disease (cGVHD)
* Received systemic therapies for cGVHD;
* Stable dose of glucocorticoids, other immunosuppressant therapy received within 2 weeks prior to screening;
* Absolute Neutrophil Count (ANC) ≥ 1.0×10 9/L ；platelet count (PLT) ≥30×10 9 /L; Hemoglobin ≥80g/L; There were no obvious abnormalities in liver and kidney function and coagulation function;
* Men and women of childbearing age agree to use contraceptive measures during the study period and within 6 months after the end of the study

Exclusion Criteria:

* Currently present or occured other malignancies within 3 years prior to first administration;
* Known or suspected active acute graft versus host disease (aGVHD);
* Presence of infection requiring treatment within 7 days prior to randomization;
* Failed allogeneic hematopoietic stem cell transplantation within 6 months or 2 prior allogeneic hematopoietic stem cell transplants;
* Use of Janus-activated kinase (JAK) inhibitors, Bruton's tyrosine kinase (BTK) inhibitors, or other, chemotherapeutic agents within 2 weeks prior to randomization;
* Has a variety of factors that affect oral medications (e.g., inability to swallow, , intestinal obstruction, etc;
* Those who have a history of psychotropic drug abuse and cannot be abstained from or have a mental disorder;
* Have any severe or uncontrolled serious illness, including but not limited to uncontrolled hypertension, heart disease, hepatitis and epilepsy that require treatment;
* Have any severe or uncontrolled serious illness, including but not limited to，uncontrolled hypertension heart disease, hepatitis and epilepsy that require treatment;
* Those who are allergic to the study drug or its components;
* Participation in other clinical trials or major surgery within 4 weeks prior to the first dose;
* Subjects judged by the investigator to be unsuitable for enrollment;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) at 24 weeks | Up to 24 weeks
  Percentage of subjects with an overall response of all evaluable organs as complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Best objective response rate (BOR) | Up to 48 weeks
  Proportion of subjects achieving CR+PR and at any time point prior to initiation of other systemic therapies for cGVHD
Duration of response (DOR) | Up to 48 weeks
  Time to first response to cGVHD disease progression, death, or initiation of any new systemic therapy for cGVHD
Failure-free survival (FFS) | Up to 48 weeks
  The time from the first dose to the time of recurrence, death, or death or increase in non-original disease or initiation of a new cGVHD systemic
Incidence rate of malignancy relapse or recurrence | Up to 48 weeks
  Proportion of subjects with recurrence date of blood system disease from the first dose
Non relapse mortality | At least 48 weeks
  From first dose to the date of death, with no recurrence of the original disease
Overall Survival (OS) | At least 48 weeks
  Time from first dose to death caused by various reasons
Adverse event rate | Up to 48 weeks
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) , evaluated according to the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0)
Severity of adverse events (AEs) | Up to 48 weeks
  Severity of all adverse medical events that occur after the subject receives the investigational drug, evaluated according to the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The 940th hospital of joint logistics support force of Chinese people's liberation army, Lanzhou, Gansu
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Tai'an Central Hospital, Taian, Shangdong
  - Ruijin Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shannxi
  - Hematology Hospital of the Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Affiliated People's Hospital of Ningbo University, Ningbo, Zhejiang